CLINICAL TRIAL: NCT01129921
Title: Comparative Study of Sham Versus Mild® (Minimally Invasive Lumbar Decompression) Procedure in Patients Diagnosed With Symptomatic Moderate to Severe Lumbar Central Canal Stenosis
Brief Title: Comparative Study of Sham Versus Mild® Procedure in Patients Diagnosed With Symptomatic Lumbar Central Canal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Napa Pain Institute (Other)
Collaborators: Vertos Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Eric J. Grigsby, MD, Founder / Medical Director, Napa Pain Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol #G01
Record Dates: First submitted 2010-04-30; First posted 2010-05-25 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Lumbar Spine Stenosis Central Canal
Keywords: Lumbar Spine Stenosis; Decompression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decompression with mild® Device Kit (Active Comparator): Fluoroscopically guided percutaneous lumbar decompression using the Vertos mild® Device Kit for bone and tissue removal to decompress the targeted stenosed level(s).
  Interventions: Device: Percutaneous Lumbar Decompression
- Sham lumbar decompression (Sham Comparator): Sham procedure of fluoroscopically guided percutaneous placement of mild® Device Kit instrumentation with no removal of bone or tissue.
  Interventions: Device: Sham lumbar decompression

INTERVENTIONS:
Device: Percutaneous Lumbar Decompression — Fluoroscopic percutaneous lumbar decompression of the central spinal canal
  Other Names: mild® Device Kit percutaneous decompression
  Arms: Decompression with mild® Device Kit
Device: Sham lumbar decompression — Sham fluoroscopic percutaneous lumbar decompression with no bone or tissue removal.
  Arms: Sham lumbar decompression

SUMMARY:
This is a single-center, randomized, prospective, double-blind, clinical study to assess the clinical application and outcomes with mild® devices versus sham in patients with symptomatic moderate to severe central canal spinal stenosis. Sham patients were eligible to choose to cross-over and have the actual decompression procedure after week 6 exam.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and lumbar spine stenosis (LSS) primarily caused by dorsal element hypertrophy.
* Prior failure of conservative therapy and Oswestry Disability Index (ODI) Score of >20%.
* Radiologic evidence of LSS, ligamentum flavum hypertrophy (typically > 2.5mm)confirmed by pre op MRI and/or CT.
* Central canal cross sectional area clearly reduced per MRI/CT report.
* If present, anterior listhesis ≤ 5.0mm (preferred) and stable.
* Able to walk at least 10 feet unaided before being limited by pain.
* Available to complete 26 weeks of follow-up.
* A signed Informed consent Form is obtained from the subject.
* Adults at least 18 years of age.

Exclusion Criteria:

* Prior surgery at intended treatment level.
* History of recent spinal fractures with concurrent pain symptoms as determined by the Investigator.
* Disabling back or leg pain from causes other than LSS (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
* Disk protrusion or osteophyte formation severe enough to confound study outcome.
* Facet hypertrophy severe enough to confound study outcome.
* Bleeding disorders and/or current use of anti-coagulants.
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory (NSAID) within five days of treatment.
* Epidural steroid administration within prior 3 weeks(of procedure or sham)
* Inability of the subject to lie prone for any reason with anesthesia support (e.g. chronic obstructive pulmonary disease (COPD), obesity, etc.).
* Metabolic wound healing pathologies deemed by Investigator to compromise study outcome.
* Dementia and/or inability to give informed consent.
* Pregnancy and/or breastfeeding.
* On Workman's Compensation or considering litigation associated with back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grigsby, MD, Principal Investigator — Napa Pain Institute
Locations (1):
- Napa Pain Institute, Napa, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred 4-19-10 to 7-28-10
Pre-assignment Details: Randomization occurred in blocks of four. After Week 6 post-treatment and prior to Week 12, Sham arm participants were allowed to have the mild decompression procedure with bone and tissue removal if they chose to have it.
Groups:
- Percutaneous Decompression Procedure Only: Group 1: Percutaneous decompression procedure with removal of bone and tissue using the mild device kit
- Sham Then Percutaneous Decompression With Mild: Group 2: After post-treatment Week 6 and prior to Week 12, patients in Sham procedure arm were allowed to participate in the active (mild procedure) study arm in which bone and tissue were removed using the mild device kit.
Period: Prior to Sham Cross-over, 6-12 Weeks
Arm/Group | Percutaneous Decompression Procedure Only | Sham Then Percutaneous Decompression With Mild
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: After Sham Cross-over to Mild, One Year
Arm/Group | Percutaneous Decompression Procedure Only | Sham Then Percutaneous Decompression With Mild
Started | 20 | 20
Completed | 18 (All 20 completed Wk 6-12 Intent to Treat analysis. Eighteen reported Year 1 outcomes.) | 13 (All 20 completed Wk 6-12 Intent to Treat analysis prior to x-over. After x-over 13 reported Year 1.)
Not Completed | 2 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — pancreatic cancer progressed | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT analysis includes all patients at weeks 6 to 12 post-treatment. Year 1 cohort analysis includes the 18 mild patients who reported outcomes at Year 1 and the 13 sham patients who reported outcomes at Year 1 after cross-over to mild.
Groups:
- Mild Procedure: Group 1: mild percutaneous decompression with removal of bone and tissue
- Sham Procedure: Group 2: sham decompression with trocar placement and no bone or tissue removal
- Total: Total of all reporting groups
Arm/Group | Mild Procedure | Sham Procedure | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 13 | 12 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.8) | 67 (12.5) | 66.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) <=4
Description: Using VAS, pain is measured on a 0 to 10 point scale where 0 represents no pain and 10 indicates severe pain. A post-treatment score of 4 points is the accepted threshold between a "mild" pain score of 1-3 points and a "moderate to severe" pain score of 5 to 10 points which represents debilitating pain that would qualify the patient for a different or additional treatment option. All patients in each arm who reported a pain score of 4 or less at six to twelve weeks post-treatment are reported below.
Time Frame: Week 6 to 12 prior to cross-over
Population: All 40 participants (20 in each arm) reported VAS at six weeks to twelve weeks post-treatment. All measurements for the sham group occurred prior to cross-over to the mild procedure. Patients with scores of 4 or less in each study group are reported below. This is Intent to Treat (ITT)analysis.
Measure: Number; unit: participants
Groups:
- Mild Procedure Group 1: Percutaneous decompression with removal of small amounts of bone and tissue to relieve stenosis.
- Sham Procedure Group 2 Prior to Cross-over: Sham placement of trocar as in percutaneous decompression, with no bone or tissue removal.
Arm/Group | Mild Procedure Group 1 | Sham Procedure Group 2 Prior to Cross-over
Number analyzed (Participants) | 20 | 20
participants | 11 (2.1) | 2 (1.8)

2. Primary Outcome: Visual Analog Scale (VAS) <=4
Description: VAS as measured on a 10-point scale. A score of 4 or less after treatment is considered favorable, as it indicates pain is less than the "moderate to severe" categories represented by scores of 5 to 10. All patients in each arm who reported a pain score of 4 or less at Week 6-12 and Year 1 are reported below.
Time Frame: Week 6 to 12 & Year One After Sham to mild x-over
Population: Patients who reported Year 1 outcomes are reported at Week 6-12 and at Year 1. All findings reported below for the Sham group are after cross-over to mild.
Measure: Number; unit: participants
Groups:
- Mild Group 1 Year-1 Cohort: Group 1: Percutaneous decompression procedure with removal of bone and tissue using the mild device kit
- Sham Group 2 Year-1 Cohort After X-over to Mild: Group 2: After post-treatment Week 6 and prior to Week 12, patients in Sham procedure arm were allowed to participate in the active (mild procedure) study arm in which bone and tissue were removed using the mild device kit.
Arm/Group | Mild Group 1 Year-1 Cohort | Sham Group 2 Year-1 Cohort After X-over to Mild
Number analyzed (Participants) | 18 | 13
participants
  Week 6-12 | 9 | 5
  Year 1 | 12 | 5

3. Primary Outcome: Visual Analog Scale (VAS) Mean Improvement
Description: VAS ten point scale where 0 = no pain and 10 represents worst pain imaginable. Mean improvement of two or more points is considered clinically relevant. The mean improvement from Baseline to Year-1 is presented below for the two treatment groups.
Time Frame: Baseline and Year 1
Population: All patients who reported Year-1 outcomes (Year-1 Cohort) were analyzed. The Sham Year-1 cohort represent those original Sham patients who crossed over from Sham to the mild procedure and were then followed for one year.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Percutaneous Decompression Procedure Only: Mild Group 1 Year-1 Cohort: Percutaneous decompression procedure with removal of bone and tissue using the mild device kit
- Sham Then Percutaneous Decompression With Mild: Sham Group 2 Year-1 Cohort: After cross-over to the active mild procedure study arm in which bone and tissue were removed using the mild device kit.
Arm/Group | Percutaneous Decompression Procedure Only | Sham Then Percutaneous Decompression With Mild
Number analyzed (Participants) | 18 | 13
units on a scale | 2.3 (2.1) | 2.2 (2.9)

ADVERSE EVENTS:
Time Frame: Throughout study to Year One
Groups:
- Mild Procedure: percutaneous decompression with bone and tissue removal
- Sham Procedure With Optional Crossover to Mild Post-unblinding: Sham procedure includes percutaneous trocar placement with no tissue or bone removal.
Arm/Group | Mild Procedure | Sham Procedure With Optional Crossover to Mild Post-unblinding
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This was a small series with challenging patient retention, particularly in the sham arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No